CLINICAL TRIAL: NCT04684706
Title: A Within Study on the Effects of L-dlPFC Activation Through iTBS in Refractory Depression
Brief Title: Compressed Intermittent Theta Burst Stimulation
Acronym: ciTBS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Yvette Sheline, Director, Center for Neuromodulation in Depression and Stress (CNDS), University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 834723
Record Dates: First submitted 2020-10-12; First posted 2020-12-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Treatment Resistant Depression
Keywords: TMS; fMRI
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Compressed iTBS schedule (Other): Stimulation 3-pulse 50-Hz bursts at 5-Hz for 2-s trains, with trains every 10 s, for 10 minutes, 10 times a day, for 5 consecutive days.
  Interventions: Device: intermittent Theta Burst Stimulation

INTERVENTIONS:
Device: intermittent Theta Burst Stimulation — The present study will utilize TMS dosage of iTBS of 18 000 pulses a day for 5 consecutive days.

SUMMARY:
In this proposal the investigators will use an accelerated TMS protocol that concentrates the magnetic stimulation that would usually occur over 6 weeks into 10 treatment sessions per days, for 5 consecutive days in patient with treatment-refractory depression. This protocol will build on a previously published study demonstrating clinical efficacy of intermittent theta-burst stimulation (iTBS) on left dorsolateral prefrontal cortex (L-dlPFC) in a treatment refractory population.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a disabling mental disorder with a lifetime prevalence of up to16% . Approximately 30% of MDD patients suffer treatment resistant depression (TRD), with at least 2 failed adequate trials of pharmacotherapy. Repetitive transcranial magnetic stimulation (rTMS) has been shown to be a safe treatment for TRD, yet the standard clinical technique for using it as treatment depressive disorders is associated with limited efficacy to date. Among the potential causes of limited efficacy have been the scalp based targeting technique that is currently the most common targeting method rather than techniques that incorporate functional magnetic resonance imaging (fMRI) neuronavigation, which have been shown to have greater efficacy. Image guided TMS can target specific functional brain networks with greater resolution that takes into account individual differences in brain anatomy.

Another technique for improving treatment efficacy, shown to modulate cortical excitability, may be the application of intermittent theta-burst stimulation in regular intervals, which has been shown to be no different than a longer-in-time application of rTMS. Paired with the evidence that iTBS has produced significant antidepressant responses in severely depressed individuals, and that relapse in depressive states predicts diminished efficacy of treatment as well as increased quantity of TBS pulses to have a beneficial effect, these recent iTBS findings suggest that iTBS may offer a valid treatment alternative to options that have proven otherwise ineffective in treating TRD. Therefore, the investigators aim to administer iTBS to severely-depressed participant in a shorter amount of time, in order to improve their antidepressant outcome.

Significance: This protocol builds on different notions:

1. iTBS is not different in treatment outcome than rTMS while applying the same amount of pulses in shorter amount of time;
2. The degree of treatment resistance is indicative of iTBS quantity needed to obtain an antidepressant treatment
3. Repeated iTBS produces a significant effect in treating refractory depression
4. Decreasing the interval between iTBS applications enhanced positive treatment outcomes.

Therefore, the compression of iTBS pulses with shorter intervals between sessions is hypothesized to have an increased beneficial effect on individuals affected by treatment-resistant depression.

ELIGIBILITY:
Inclusion Criteria:

* Gender, inclusive
* 18 - 70 years of age
* Meets Diagnostic and Statistical Manual of Mental Disorders criteria for primary diagnosis of MDD
* Patients must be fluent in English
* Participants must have the ability to provide consent
* Montgomery Asberg Depression Rating Scale score ≥20
* Failed 2+ prior treatments (treatment-refractory)
* May be on current anti-depressant medication at the discretion of PI, if not exceeding doses that would make TMS an increased risk

Exclusion Criteria:

* Pregnancy (Female participants)
* MRI contraindication
* Medical condition that interferes with the collection or interpretation of MRI data
* Implanted devices such as: aneurysm clip or cardiac pacemaker
* Diagnosis of stroke, epilepsy, or other neurological disorders interfering with treatment at PI discretion
* Any factor the investigator believe may affect participant safety or compliance (ex: ≥100 miles from clinic)
* Current alcohol or substance use disorder in last 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptoms Change | 2 Weeks
  Depressive symptoms will be measured before and after treatment by means of the clinician-administered Montgomery Asberg Depression Rating Scale (MADRS) (0-60, lower scores indicate lower depressive symptoms) and the self report Beck Depression Inventory (BDI II) (0-30, lower scores indicate lower depressive symptoms). Change will be measured by comparing measurements pre- and post- on the same measures. The bigger the change, the bigger the reduction in depressive symptoms.

SECONDARY OUTCOMES:
Self report Symptom Change | 2 weeks
  Depressive symptoms will be measured before and after treatment by means of the self report Beck Depression Inventory (BDI II) (0-30, lower scores indicate lower depressive symptoms). Change will be measured by comparing measurements pre- and post- on the same measures. The bigger the change, the bigger the reduction in depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Sheline, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Department of Interventional Psychiatry, University of California San Diego, La Jolla, California
  - Center for Neuromodulation in Depression and Stress, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No